CLINICAL TRIAL: NCT06841939
Title: Effectiveness of Castor Oil in Preventing Formal Induction of Labour Among Pregnant Women at a Tertiary Institution in Abakaliki: A Randomized Controlled Trial.
Brief Title: Effectiveness of Castor Oil in Preventing Formal Induction of Labour in a Tertiary Institution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assumpta Nnenna Nweke (Other Government)
Responsible Party: Sponsor-Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Organization: Federal Teaching Hospital Abakaliki (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AEFUTHA/REC/VOL.3/2020/015
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Castor Oil; Prolonged Pregnancy
Keywords: Castor oil; Induction of labour; Prolonged pregnancy
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Castor Oil; Water

STUDY DESIGN:
Intervention Model Description: open label clinical superiority randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Castor oil (Experimental): Participants recruited into this group had vaginal examinations conducted and it was confirmed that they were not in labour, Bishop's score was then documented. They were counselled to take 30 ml of castor oil under direct observation by the researcher and the time and date of administration documented. The participants' phone numbers and addresses were also recorded. Participants who fail to achieve labour within 24 hours had a repeat dose of 30 ml of castor oil.
  Interventions: Other: castor oil
- Water (Placebo Comparator): Participants recruited into this group had vaginal examinations conducted and it was confirmed that they were not in labour, Bishop's score was then documented. They were counselled to take 30 ml of water under direct observation by the researcher and the time and date of administration documented. The participants' phone numbers and addresses were also recorded. Participants who fail to achieve labour within 24 hours had a repeat dose of 30 ml of water.
  Interventions: Other: Water

INTERVENTIONS:
Other: castor oil — Participants recruited into this group had vaginal examinations conducted and it was confirmed that they were not in labour, Bishop's score was then documented. They were counselled to take 30 ml of castor oil under direct observation by the researcher and the time and date of administration documented. The participants' phone numbers and addresses were also recorded. Participants who fail to achieve labour within 24 hours had a repeat dose of 30 ml of castor oil.
  Arms: Castor oil
Other: Water — Participants recruited into this group had vaginal examinations conducted and it was confirmed that they were not in labour, Bishop's score was then documented. They were counselled to take 30 ml of water under direct observation by the researcher and the time and date of administration documented. The participants' phone numbers and addresses were also recorded. Participants who fail to achieve labour within 24 hours had a repeat dose of 30 ml of water.
  Arms: Water

SUMMARY:
This study demonstrated that castor oil was effective in reducing the need for formal induction of labour and the administration-delivery interval with minimal maternal side-effects, at an initial dose of 30ml and single repeat dose of 30ml.

DETAILED DESCRIPTION:
Background: Pregnancy extending beyond 42 week is attended by maternal and perinatal complication including death. It is the commonest reason for induction of labour. Various agents have been used to induce labour but it is not without maternal and fetal side effects. Alternative agents such as castor oil have been widely used in clinical practice for induction of labour without any concrete evidence of effectiveness.

Objective: To evaluate the effectiveness of castor oil in the prevention of formal induction of labour amongst pregnant mothers at Alex Ekwueme Federal University Teaching Hospital Abakaliki as well as to evaluate the possible maternal and fetal/ neonatal effects.

Methods: This was a randomized controlled trial among pregnant women at Alex Ekwueme Federal University Teaching Hospital Abakaliki to verify the effectiveness of castor oil in the prevention of formal induction of labour at gestational ages between 41weeks and 0 days and 41 weeks and 2 days. One arm received 30ml of castor oil (Group A) and the other arm received 30ml of water (Group B). These doses were repeated once more after 24 hours if the patients failed to enter spontaneous labour. The data obtained was analyzed using IBM SPSS software (version 24, Chicago II, USA) and the intention to treat concept. A difference with a P value of ≤ 0.05 was taken to be of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of 41weeks+0day to 41weeks+2days
2. Pregnancies with cephalic presenting fetuses
3. Pregnant women with singleton fetus
4. Absence of contraindications to vaginal delivery
5. Absence of uterine contraction
6. Bishop score ≤ 5
7. Ultrasound confirmed GA in early pregnancy

Exclusion Criteria:

1. Pregnant women in latent phase of labour
2. Preterm or term premature rupture of membrane
3. Antepartum haemorrhage
4. Previous Caesarean section and myomectomy
5. Multiple gestation
6. Medical disorders of pregnancy
7. Unsure date

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
formal Induction of labour | 24 hours
  proportion of women who had formal induction of labour

CONTACTS AND LOCATIONS:
Overall Officials: Assumpta N Nweke, MBBSMBBS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital Abakaliki Ebonyi State
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No